CLINICAL TRIAL: NCT00958529
Title: Effect of Two Doses of Inulin Products on Gastrointestinal Tolerance
Brief Title: Gastrointestinal Toleration of Inulin Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Cargill (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0805M32121
Record Dates: First submitted 2009-08-12; First posted 2009-08-13 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Healthy
Keywords: fiber; inulin; gastrointestinal tolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- inulin (Experimental): 0, 5, 10 g inulin
  Interventions: Dietary Supplement: Inulin Fiber Supplement

INTERVENTIONS:
Dietary Supplement: Inulin Fiber Supplement — Orange juice fortified with 0, 5g, and 10g of 2 inulin products

SUMMARY:
The intake of inulin products has been linked to multiple health benefits which has lead to inulin fortification in food products.

The investigators hypothesis that doses of up to 10 grams of inulin products should be well tolerated and not result in a significant increase in gastrointestinal symptoms.

DETAILED DESCRIPTION:
0, 5, and 10 grams of inulin

ELIGIBILITY:
Inclusion Criteria:

* english speaking
* healthy men and women
* 18 and 60 years of age
* non-smoking
* non-dieting
* BMI less than 30
* standard diet consisting of no more than 15 grams fiber
* not taking medications

Exclusion Criteria:

* BMI more than 30
* CVD
* Diabetes Mellitus
* cancer in prior 5 years
* renal or hepatic disease
* bacterial infection in past 2 weeks
* more than 5 kg weight loss in past 3 months
* history of drug or alcohol abuse in past 6 months
* use of weight loss, lipid-lowering, anti-hypertensive, or anti- inflammatory medications
* concurrent or recent intervention study participation
* consumption of laxatives
* history of gastrointestinal disorders
* food allergies
* pregnant or lactating women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2008-08; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal Tolerance Score | Aug 2008 thru Oct 2008

CONTACTS AND LOCATIONS:
Overall Officials: Joanne L Slavin, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota: Nutrition and Food Science Department, Minneapolis, Minnesota, United States